CLINICAL TRIAL: NCT00594373
Title: Effect of Repeated Applications of Tenofovir Gel on Mucosal Mediators of Immunity and Intrinsic Antimicrobial Activity of Cervicovaginal Secretions in Women at Low Risk for HIV-1 Infection
Brief Title: Interventional Study of Mucosal and Antimicrobial Responses to Repeated Vaginal Applications of Tenofovir Gel in HIV Uninfected Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TFV 010; 10443 (Registry Identifier: DAIDS ES); U01AI069551 (NIH)
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Microbicide; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — hexadecyloxypropyl 9-(2-(phosphonomethoxy)propyl)adenine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Application of 1% tenofovir gel for 14 consecutive days between menses
  Interventions: Drug: Tenofovir gel
- 2 (Placebo Comparator): Application of 1% tenofovir placebo gel for 14 consecutive days between menses
  Interventions: Drug: Tenofovir gel placebo

INTERVENTIONS:
Drug: Tenofovir gel — 1 gm/100 ml of 1% tenofovir gel vaginally daily
  Other Names: TFV; 9-(2-[Phosphonomethoxy]propyl)adenine
  Arms: 1
Drug: Tenofovir gel placebo — 1 gm/100 ml of placebo gel vaginally daily
  Arms: 2

SUMMARY:
Topical microbicides, substances that kill microbes, are being studied to prevent sexual transmission of HIV and other disease-causing agents. In the future, topical microbicides may be applied vaginally to prevent both acquisition and transmission of HIV and other sexually transmitted infections (STIs). The purpose of this study is to assess whether there is a measurable response to daily applications of a topical microbicide, 1% tenofovir gel, in women at low risk for HIV infection.

DETAILED DESCRIPTION:
A new approach to HIV prevention currently being studied is the use of topical microbicides. This study will measure the mucosal response to daily intravaginal applications of 1% tenofovir gel versus placebo in two groups of women at low risk for HIV infection.

The duration of this study for each participant is 21 days. Study participants will be randomly assigned to one of two study groups. Group 1 participants will apply 1% tenofovir gel daily for 14 consecutive days between menses. Group 2 participants will apply placebo gel for 14 consecutive days between menses.

Study visits will occur on Days 3, 7, 14, and 21. Study entry will occur 2 to 6 days following the menses and within 30 days of screening. Medical and sexual history, a pelvic exam, cervicovaginal lavage sample collection, blood collection, vaginal pH testing, STI testing, and adverse effect reporting will occur at all visits. All participants will be asked to complete a diary throughout the study; this diary will be reviewed at all study visits. A Pap smear will be obtained at screening if documentation of a negative Pap smear result within the last year is not available.

ELIGIBILITY:
Inclusion Criteria:

* Normal menstrual history with regular cycles and with a minimum of 21 days between menses
* Sexually abstinent or in a stable, mutually monogamous relationship with a partner who is HIV uninfected
* Agree to abstain from sexual intercourse and to not use vaginal products within 48 hours of study entry and for the duration of the study

Exclusion Criteria:

* HIV infected
* Sexually transmitted infection within 6 months of study entry
* Use of nontherapeutic intravenous drugs within 12 months of study entry
* Menopausal
* Currently using hormonal contraception or have used hormonal contraception within 2 months of study entry
* Menstruating at screening or enrollment visits
* Positive urine culture
* Positive chlamydia, gonorrhea, or trichomonas result at screening
* Abnormal Pap smear
* Clinically detectable genital abnormality. More information on this criterion can be found in the protocol.
* History of toxic shock syndrome or a history of symptoms suggesting toxic shock syndrome
* History of intermenstrual bleeding within 3 months of study entry
* Previous gynecologic surgery or have received treatment for syphilis, genital herpes, chlamydia, gonorrhea, trichomonas, or genital warts within 6 months of study entry
* Received treatment for Candida, bacterial vaginosis, or urinary tract infection within 1 month of study entry
* Have douched or used vaginal products, including lubricants, feminine hygiene products, vaginal drying agents, and sex toys within 48 hours of study entry
* Acute or chronic hepatitis B virus infection
* Liver or kidney abnormalities
* Oral antibiotics within 7 days of study entry
* Pregnant, less than 6 months postpartum, or breastfeeding

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Changes in cytokines, chemokines, and other mediators of innate immunity through examination of cervicovaginal secretions | At Days 3, 7, 14, and 21

SECONDARY OUTCOMES:
Changes in antimicrobial activity of cervicovaginal secretions | At Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Marla Keller, MD, Principal Investigator — Albert Einstein College of Medicine; Betsy Herold, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine - East Campus GCRC (Herold) Non-Network CRS, The Bronx, New York, United States

REFERENCES:
- [Background] Bateman C. Tenofovir gel--the new HIV prevention 'banker'? S Afr Med J. 2007 Jul;97(7):496, 498. No abstract available. PMID 17805450
- [Background] Mayer KH, Maslankowski LA, Gai F, El-Sadr WM, Justman J, Kwiecien A, Masse B, Eshleman SH, Hendrix C, Morrow K, Rooney JF, Soto-Torres L; HPTN 050 Protocol Team. Safety and tolerability of tenofovir vaginal gel in abstinent and sexually active HIV-infected and uninfected women. AIDS. 2006 Feb 28;20(4):543-51. doi: 10.1097/01.aids.0000210608.70762.c3. PMID 16470118
- [Derived] Keller MJ, Madan RP, Torres NM, Fazzari MJ, Cho S, Kalyoussef S, Shust G, Mesquita PM, Louissaint N, Chen J, Cohen HW, Diament EC, Lee AC, Soto-Torres L, Hendrix CW, Herold BC. A randomized trial to assess anti-HIV activity in female genital tract secretions and soluble mucosal immunity following application of 1% tenofovir gel. PLoS One. 2011 Jan 25;6(1):e16475. doi: 10.1371/journal.pone.0016475. PMID 21283552